CLINICAL TRIAL: NCT06707883
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II Clinical Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of TQC2731 Injection in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease
Brief Title: A Clinical Study of TQC2731 Injection in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Chia Tai Tianqing Pharmaceutical Technology Development Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQC2731-II-04
Record Dates: First submitted 2024-11-25; First posted 2024-11-27 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQC2731 injection (Experimental): TQC2731 injection, 28days as a treatment cycle.
  Interventions: Drug: TQC2731 injection
- TQC2731 Placebo (Placebo Comparator): TQC2731 Placebo, 28days as a treatment cycle.
  Interventions: Drug: TQC2731 Placebo

INTERVENTIONS:
Drug: TQC2731 injection — TQC2731 injection is a monoclonal antibody that blocks thymic stromal lymphopoietin (TSLP)
  Arms: TQC2731 injection
Drug: TQC2731 Placebo — TQC2731 Placebo without drug substance.
  Arms: TQC2731 Placebo

SUMMARY:
To evaluate the efficacy and safety of TQC2731 injection in patients with moderate to severe chronic obstructive pulmonary disease.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide written informed consent and comply with the study protocol;
* Participant must be ≥40 to ≤80 years of age at the time of signing informed consent.
* Participants with a physician diagnosis of Chronic Obstructive Pulmonary Disease(COPD) and a history of COPD ≥12 months with medical records or related records at the time of screening;
* Post-bronchodilator FEV1/Forced vital capacity (FVC)<0.70 and post-bronchodilator FEV1 % predicted ≥20% and < 80% during screening.
* Modified Medical Research Council (mMRC) Dyspnea Scale grade≥2 during screening.
* Background triple therapy (ICS+long-acting beta-agonists (LABA)+LAMA) for at least 3 months with a stable dose for at least 1 month prior to randomization; Double therapy allowed if ICS is contraindicated.
* With a history of acute exacerbation of ≥2 moderate or ≥1 severe within the previous 12 months prior to screening. Multiple acute exacerbation events with an interval of less than 14 days are counted as one.

Exclusion Criteria:

* COPD with asthma;
* Subjects with active pulmonary diseases other than COPD assessed by the investigator.
* Moderate to severe Acute exacerbations of chronic obstructive pulmonary disease (AECOPD) occurred within 4 weeks prior to screening or during screening;
* History of lung transplantation;
* Previous use of TQC2731.
* Diagnosis of alpha-1 anti-trypsin deficiency;
* History of lung volume reduction surgery or pneumonectomy within 6 months prior to randomization, or planned lung volume reduction surgery during the study period;
* Positive hepatitis B surface antigen, or hepatitis C virus antibody, or syphilis antibody.
* Diagnosis of immunodeficiency, including but not limited to HIV infection;
* Infection requiring systemic therapy within 2 weeks prior to randomization.
* Starting rehabilitation within 4 weeks prior to randomization, or planned rehabilitation during the study period;
* Treatment with oxygen of more than 12 hours per day.
* Heart failure New York Heart Association (NYHA) class III or IV during the screening period.
* History of malignancy within 5 years prior to screening, excluding cervical carcinoma in situ, ductal carcinoma in situ, etc.
* Pregnancy or breastfeeding.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2024-12-31 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Annual rate of acute COPD exacerbation | Baseline to week 24
  Annualized rate of moderate or severe COPD exacerbations over the 24-week treatment period compared to placebo

SECONDARY OUTCOMES:
Change in pre-bronchodilator forced expiratory volume (FEV1) | Baseline to week 24
  Change in pre-bronchodilator FEV1 from baseline to week 24 compared to placebo.
Annual rate of acute COPD exacerbation | Baseline to week 52
  Annualized rate of moderate COPD exacerbations over the 52-week treatment period compared to placebo.
Improvement in St. George's Respiratory Questionnaire (SGRQ) | Baseline to week 52
  Proportion of patients with SGRQ improvement ≥4 points at Week 52
Change in SGRQ | Baseline to week 52
  Change from baseline to Week 52 in SGRQ total score compared to placebo
Change in pre-bronchodilator FEV1 | Baseline to week 52
  Change in pre-bronchodilator FEV1 from baseline to week 52 compared to placebo.
Annual rate of acute COPD exacerbation | Baseline to week 52
  Annualized rate of severe COPD exacerbations over the 52-week treatment period compared to placebo.
Change in post-bronchodilator FEV1 | Baseline to week 24 and 52
  Change in post-bronchodilator FEV1 from baseline to week 24 and 52 compared to placebo.
Change in EXACT | Baseline to week 52
  Change from baseline to Week 52 in EXACT total score compared to placebo.
Adverse Events (AE) and Serious Adverse Events (SAE) | Baseline to 64 weeks
  The incidence and severity of AE and SAE, as well as abnormal laboratory examination index.
Anti-drug antibodies (ADA) | Baseline through week 52
  Incidence of ADA.
Immunoglobulin E (IgE) | Baseline to 52 weeks
  Changes in IgE levels in peripheral blood.
Fractional exhaled nitric oxide (FeNO) | Baseline to 52 weeks
  Changes in FeNO.

CONTACTS AND LOCATIONS:
Locations (60):
- China (60):
  - The First People's Hospital of Chuzhou, Chuzhou, Anhui
  - The second hospital of ANHUI medical university, Hefei, Anhui
  - Huainan Dongfang Hospital Group General Hospital, Huainan, Anhui
  - Capital Medical University Beijing Chaoyang Hospital, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Shunde Hospital Of Southern Medical University, Foshan, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Jiangmen Central Hospital, Jiangmen, Guangdong
  - Affiliated Qingyuan Hospital,Guangzhou Medical University,Qingyuan People's Hospital, Qingyuan, Guangdong
  - Zhongshan City People's Hospital, Zhongshan, Guangdong
  - Nanxishan Hospital of Guangxi Zhuang Autonomous, Guilin, Guangxi
  - The First People' Hospital Of YuLin, Yulin, Guangxi
  - Zunyi Medical University Affiliated Hospital, Zunyi, Guizhou
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Jiaozuo Second People's Hospital, Jiaozuo, Henan
  - The First Affiliated Hospital of Henan University of Science & Technology, Luoyang, Henan
  - Puyang Oilfield General Hospital, Puyang, Henan
  - Henan Chest Hospital, Zhengzhou, Henan
  - Jianghan University Affiliated Hospital (Wuhan Sixth Hospital), Wuhan, Hubei
  - Wuhan Central Hospital, Wuhan, Hubei
  - Yichang Central People's Hospital, Yichang, Hubei
  - Changsha First Hospital, Changsha, Hunan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangtan County People's Hospital, Xiangtan, Hunan
  - Xiangya Hospital Zhuzhou Central South University, Zhuzhou, Hunan
  - Inner Mongolia Autonomous Region People's Hospital, Hohhot, Inner Mongolia
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - Jiangyin Hospital of Traditional Chinese Medicine, Jiangyin, Jiangsu
  - The Fifth People's Hospital of Wuxi, Wuxi, Jiangsu
  - Yixing People'S Hospital, Wuxi, Jiangsu
  - XuZhou Central Hospital, Xuzhou, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - Xinyu People'S Hospital, Xinyu, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - General Hospital of Anshan Iron and Steel Group Corporation, Anshan, Liaoning
  - Benxi Central Hospital, Benxi, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Heze Municipal Hospital, Heze, Shandong
  - Linyi People's Hospital, Linyi, Shandong
  - Qingdao Municipal Hospital, Qingdao, Shandong
  - Weifang NO.2 People' Hospital, Weifang, Shandong
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Shanghai JiaoTong University of medicine Ruijin Hospital, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Affiliated Hospital Of ChengDu University, Chengdu, Sichuan
  - Guangyuan Central Hospital, Guangyuan, Sichuan
  - Leshan People's Hospital, Leshan, Sichuan
  - Meishan People's Hospital, Meishan, Sichuan
  - Suining Central Hospital, Suining, Sichuan
  - General Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - The Fourth Central Hospital of Tianjin, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Shihezi University, Shihezi, Xinjiang
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Jiaxing Second Hospital, Jiaxing, Zhejiang
  - Taizhou Central Hospital Central Hospital, Taizhou, Zhejiang
  - The 2th School of Medicine ,WMU/The 2th affiliated Hospital and Yuying Children's Hospital of WMU, Wenzhou, Zhejiang